CLINICAL TRIAL: NCT03054779
Title: Canola Oil Multi-center Intervention Trial II (COMIT II): Effects of Oleic Acid Enriched and Regular Canola Oil on Body Composition and Lipid Metabolism in Participants With Metabolic Syndrome Risk Factors
Brief Title: Canola Oil Multi-center Intervention Trial II
Acronym: COMITII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Canola Council of Canada (Other); University of Manitoba (Other); Laval University (Other); Unity Health Toronto (Other); St. Boniface Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: PKE COMIT II
Record Dates: First submitted 2015-04-28; First posted 2017-02-16 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease; Metabolic Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome | interventions — Rapeseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Canola oil (Experimental): regular canola oil
  Interventions: Other: Canola Oil
- High oleic acid canola oil (Experimental): high stability/high oleic canola oil
  Interventions: Other: High oleic acid canola oil
- Western diet oil combination (Active Comparator): a typical "Western diet" fat intake comprised of 11% MUFA, 11% PUFA (9% omega-6 fatty acids and 2% omega-3 fatty acids), and 13% SFA
  Interventions: Other: Western diet oil combination

INTERVENTIONS:
Other: Canola Oil — Regular canola oil will be iso-calorically incorporated into fruit smoothies made with milk and consumed twice daily.
  Arms: Canola oil
Other: High oleic acid canola oil — High oleic acid canola oil will be iso-calorically incorporated into fruit smoothies made with milk and consumed twice daily.
  Arms: High oleic acid canola oil
Other: Western diet oil combination — A typical "Western diet" fat intake as a control treatment, comprised of 11% MUFA, 11% PUFA (9% omega-6 fatty acids and 2% omega-3 fatty acids), and 13% SFA, will be iso-calorically incorporated into fruit smoothies made with milk and consumed twice daily
  Arms: Western diet oil combination

SUMMARY:
Building on the findings from the investigators previous study, COMIT I, the purpose of the COMIT II study is to supplement the DEXA measurement of body composition with a supplementary DEXA measurement of visceral adipose tissue and to specifically target the impact of oleic acid consumption on body composition as the primary objective. COMIT II also will include analysis of fatty acid ethanolamines (FAEs) and their precursors to elucidate the mechanisms by which canola oil may be modifying body composition, measurement of endothelial function, inflammatory, adiposity and insulin sensitivity biomarkers, and genetic analyses.

ELIGIBILITY:
Inclusion Criteria:

* waist circumference ≥94 cm for men and ≥80 cm for women
* Elevated triglycerides - ≥150 mg/dL and ≤ 400 mg/dL
* Reduced HDL - < 40 mg/dL for men and < 50 mg/dL for women
* Fasting glucose - ≥ 100 mg/dl and ≤ 126 mg/dL
* Elevated blood pressure - systolic ≥130 and/or diastolic ≥85 mm HG [Unmedicated participants - upper limit of Stage 1 Hypertension: systolic < 160 and/or diastolic <100 mm HG and participants must be free of end stage/target organ disease symptoms] [BP medicated participants: acceptable as long as individuals meet the specified blood pressure range of <140/90 mmHg, and have been stable for at least 6 months]

Exclusion Criteria:

* Individuals with thyroid**, kidney, or liver disease [Individuals with thyroid disease whose blood values are within normal limits and that have been stable (on medication) for the past 6 months are considered eligible]
* Individuals with diabetes mellitus
* Smokers
* Individuals consuming >14 alcoholic beverages per week
* Individuals taking lipid lowering medication (ex: cholestyramine, colestipol, niacin, cloribrate, gemfibrozil, probucol, HMG CoA reductase inhibitors) for at least the last 3 months
* Pregnancy or lactation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Body composition | 1 year 6 months
  Will be measured using DXA
Plasma lipids | 1 year 6 months
Flow mediated dilation (FMD) for endothelial function | 1 year 6 months
Lipoprotein subclasses | 1 year 6 months
Inflammatory markers | 1 year 6 months
Lipid Peroxidation | 1 year 6 months

SECONDARY OUTCOMES:
Assessment of fatty acid inter-conversion and synthesis using stable isotope tracers | 1 year 6 months
Genetic analysis to evaluate the association between FADS 1 and FADS 2 mRNA and protein expression in peripheral blood mononuclear blood cells (PBMCs) | 1 year 6 months
Physical activity level | 1 year 6 months
  Will be assessed using an Actigraph GT3X+ activity monitor to be worn for 1 week at the end of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States